CLINICAL TRIAL: NCT04102878
Title: Comparative Study of Transconjunctival vs. Transcutaneous Routes for Administration of Local Anaesthesia in Oculoplastic Surgery
Brief Title: Transconjunctival vs Transcutaneous Anaesthesia in Oculoplastics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OPH0260
Record Dates: First submitted 2019-04-05; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Anesthesia, Local; Eyelid Diseases
Keywords: oculoplastic surgery
MeSH Terms: conditions — Eyelid Diseases | interventions — Anesthetics, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous anaesthetic (Active Comparator)
  Interventions: Drug: Topical Anesthetic; Procedure: Transcutaneous anaesthetic; Other: Patient comfort questionnaire; Other: Facial photograph; Procedure: Eyelid surgery
- Transconjunctival anaesthetic (Active Comparator)
  Interventions: Drug: Topical Anesthetic; Procedure: Transconjunctival anaesthetic; Procedure: Transcutaneous anaesthetic; Other: Patient comfort questionnaire; Other: Facial photograph; Procedure: Eyelid surgery

INTERVENTIONS:
Drug: Topical Anesthetic — Topical anaesthetic drops (proxymetacaine 0.5% and tetracaine 1%) applied
Procedure: Transconjunctival anaesthetic — Local anaesthetic (50/50 mixture of bupivacaine 0.5% / lidocaine 2% with adrenaline 1:200 000) administered to the eyelid via the transconjunctival route
  Arms: Transconjunctival anaesthetic
Procedure: Transcutaneous anaesthetic — Local anaesthetic (50/50 mixture of bupivacaine 0.5% / lidocaine 2% with adrenaline 1:200 000) administered to the eyelid via the transcutaneous route
Other: Patient comfort questionnaire — The patient will be asked to rate the level of pain during each local anaesthetic injection on a 0-10 scale
Other: Facial photograph — The patient will have a photograph taken following the anaesthetic injections to document the presence or absence of bruising
Procedure: Eyelid surgery — Eyelid surgery will be performed as per the plan from their preoperative appointment

SUMMARY:
Eyelid surgery is commonly performed under local anaesthesia. For many such procedures, the local anaesthetic injection may be given either transcutaneously (through the skin) or transconjunctivally (through the conjunctiva, i.e. from the inner surface of the eyelid after administration of topical anaesthetic drops). Both methods are commonly used, sometimes in combination. Currently, the choice of route is largely determined by surgeon preference, but it is not known whether one method is better or more comfortable than the other. Our study will compare the two methods of local anaesthetic administration, in terms of patient comfort during anaesthetic administration, efficacy (i.e. whether any additional anaesthetic is needed during surgery), and adverse effects (e.g. bruising, postoperative double vision).

We will recruit adult patients who are due to undergo eyelid surgery on both sides under local anaesthesia, on Miss Siah's lists at Southampton General Hospital or Lymington Hospital. Patients will receive topical anaesthetic eye drops to both eyes, followed by an injection of local anaesthetic to each eyelid. One side will be administered transcutaneously, and the other side transconjunctivally. The order be randomised. After the injections, participants will be asked to rate their pain levels during each injection on a standardised numerical scale (1-10). A photograph will also be taken, so that an independent assessor can subsequently rate the extent of any bruising. The eyelid surgery will then be performed as normal, with any need for further anaesthetic during the surgery being recorded. Patients will attend for their normal follow-up appointment afterwards and any postoperative complications will be recorded, but the study will not require any extra hospital visits. The study is sponsored by University Hospitals NHS Foundation Trust, but does not have any external funding.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing bilateral oculoplastic procedures under local anaesthesia on selected lists at Southampton General Hospital or Lymington New Forest Hospital, UK
* able to give informed consent and adhere to the study protocol

Exclusion Criteria:

* patients undergoing substantially different procedures on each eye
* patients undergoing procedures not amenable to the administration of anaesthetic via the transconjunctival route (e.g. brow lift)
* patients undergoing a first procedure on one eye and a 'redo' procedure on the fellow eye (as the presence of scar tissue on the previously operated eye is likely to affect results)
* patients having their procedure under general anaesthesia, or receiving intravenous sedation prior to the administration of local anaesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-04 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain during local anaesthetic administration | During local anaesthetic administration (2-3 minutes)
  Patient-rated pain intensity during administration of local anaesthetic via each route (transconjunctival and transcutaneous), expressed on a 0-10 scale (0 being no pain at all and 10 being the worst pain possible)

SECONDARY OUTCOMES:
Requirement for additional anaesthetic | During surgical procedure (up to 1 hour)
  Requirement (or lack thereof) for additional 'top up' anaesthetic during the eyelid surgery.
Bruising after local anaesthetic | Immediately after local anaesthetic (2-5 minutes)
  Amount of bruising visible on facial photographs taken after the anaesthetic is administered but before the eyelid surgery, rated on a numeric scale of 0-3 by an independent assessor (i.e. a member of the research team who did not perform the anaesthetic or surgery).
Other complications | During anaesthetic administration, surgery, or up until the first postoperative visit (2-3 weeks later)
  Occurrence of any other complications or adverse events potentially attributable to the administration of local anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: We Fong Siah, Principal Investigator — University Hospitals Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jawad M, Chow K, Nicholson R, Jonas A, Siah WF. Transconjunctival versus transcutaneous local anaesthetic administration for lower eyelid surgery: a randomised controlled trial. Eye (Lond). 2022 May;36(5):1094-1099. doi: 10.1038/s41433-021-01588-w. Epub 2021 Jun 11. PMID 34117385